CLINICAL TRIAL: NCT06953518
Title: An Open-Label Pilot Study of Qualia Senolytic Supplementation for the Attenuation of Systemic Inflammatory Cytokines
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qualia Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: QLS-010
Record Dates: First submitted 2025-04-16; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Inflammation
Keywords: Senolytic
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Qualia Senolytic (Active Comparator)
  Interventions: Dietary Supplement: Qualia Senolytic

INTERVENTIONS:
Dietary Supplement: Qualia Senolytic — Qualia Senolytic manufactured by Qualia Life Science

SUMMARY:
This open-label pilot study includes adults aged 45 to 79 residing in the United States. The study will last 7 days. Participants will provide blood samples via an at-home finger-prick kit at baseline and day 7 and complete electronic surveys on health indicators at baseline, and days 3 and 7. All procedures are conducted remotely, with no in-person visits, to collect real-world evidence.

DETAILED DESCRIPTION:
Objectives Within-group changes in outcomes will be compared from baseline to the end of the study period.

Primary Outcome Measures:

Biomarkers in blood, measured using the Olink Target 48 Cytokine panel:

Tumor Necrosis Factor (TNF) Interleukin-1 Beta (IL1B) Interleukin-8 (CXCL8) Vascular Endothelial Growth Factor A (VEGFA)

Secondary Outcome Measures:

Remaining biomarkers in the Olink Target 48 Cytokine panel 36-Item Short Form Health Survey (SF-36) Frailty Index for Elders (FIFE) Depression Anxiety Stress Scale-21 (DASS-21)

Side effect profile including:

Number, type, severity, causality, and outcome of adverse events or unanticipated problems

Symptoms of aging, assessed by:

Aging Male Symptom scale Aging Female Symptom scale

Participant Details:

Study Duration per Participant: 7 days Total Number of Participants: 40

ELIGIBILITY:
Inclusion Criteria:

* Provide voluntary, written, informed consent to participate in the study
* Agree to provide a valid cell phone number and are willing to receive communications through text.
* Healthy adults 45 - 79 years of age Can read and write English
* Willing to not begin taking any new supplements during the study and continue taking any supplements they are currently using regularly.
* Willing to self-administer the fingerstick test kit at home for both a baseline and post-intervention blood sample, and to complete a release form that gives NHC access to the results of these tests.
* Willing to complete questionnaires, records, and diaries associated with the study.

Exclusion Criteria:

* Women who are pregnant, breastfeeding, or planning to become pregnant during the trial
* Known food intolerances/allergy to any ingredients in the product
* Having any of the following conditions: Psychiatric conditions, neurologic disorders, endocrine disorders, cancer
* Having had a significant cardiovascular event in the past 6 months
* Taking MAO inhibitors, SSRIs, or any other psychiatric or neurological medicines
* On immunosuppressive therapy
* Individuals who were deemed incompatible with the test protocol
* Adults lacking capacity to consent

Ages: 45 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-12 (Estimated); Primary Completion 2025-05-18 (Estimated); Study Completion 2025-05-18 (Estimated)

PRIMARY OUTCOMES:
Olink Target 48 Cytokine panel - TNF, IL1B, CXCL8, VEGFA | 1 week
  Biomarkers in blood, measured using the Olink Target 48 Cytokine panel:
  Tumor Necrosis Factor (TNF) Interleukin-1 Beta (IL1B) Interleukin-8 (CXCL8) Vascular Endothelial Growth Factor A (VEGFA)

SECONDARY OUTCOMES:
Remaining biomarkers in the Olink Target 48 Cytokine panel | 1 week
36-Item Short Form Health Survey (SF-36) | 1 week
Frailty Index for Elders (FIFE) | 1 week
Depression Anxiety Stress Scale-21 (DASS-21) | 1 week
Aging Male/Female Symptom scale | 1 week
Side effect profile as measured by a custom Safety and Tolerability survey | 1 week
  Number of participants with treatment-related adverse events as assessed by a score of 3 or greater on the Safety and Tolerability survey

CONTACTS AND LOCATIONS:
Locations (1):
- Qualia Life Sciences, Carlsbad, California, United States

IPD SHARING:
Plan to Share IPD: No